CLINICAL TRIAL: NCT03413410
Title: A Multi-Center Study on the Metoprolol Optimal Dosing Pathway of Metoprolol Application in Chinese Patients With Acute Coronary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yun Dai Chen (Other)
Responsible Party: Sponsor-Investigator, Yun Dai Chen, MD, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-16-12344
Record Dates: First submitted 2018-01-11; First posted 2018-01-29 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: ACS - Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metoprolol interventional group (Experimental): This is a multi-center, prospective, open label, single-arm interventional study.
  Patients hospitalized for ACS, fulfilling all of the inclusion criteria and none of the exclusion criteria can be enrolled in this study.
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Metoprolol — Patients with acute coronary syndrome take metoprolol during hospital and after discharge in the optimal dosing pathway.

SUMMARY:
This study is to test the feasibility and tolerability of the metoprolol optimal dosing pathway by observing the percentage of patients achieving target dose followed the pathway on ACS patients during hospitalization.

DETAILED DESCRIPTION:
Acute coronary syndrome(ACS) is one of the main manifestations of cardiovascular disease and one of the main causes for hospitalization in adults.

Previous studies showed that β-receptor blockers can reduce ACS patients' cardiovascular risk in both acute phase and secondary prevention. We summarized the metoprolol optimal dosing pathway based on Chinese and foreign guidelines as well as Chinese clinical practice.

Primary endpoint is the percentage of patients achieving target dose at time of discharge.

Secondary endpoints are the mean HR & BP at discharge and during the follow up period of the Patients who have achieved target dose at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above;
* Hospitalized due to acute coronary syndrome;
* Able and willing to provide written informed consent and to comply with the study.

Exclusion Criteria:

* Cardiac shock;
* Unstable heart failure;
* Beta-agonist therapy on a continuous or intermittent basis;
* Hypotension (BP<90/60 mmHg) or bradycardia (HR<50 bpm) with symptoms;
* Sick sinus syndrome;
* Ⅱ~Ⅲ atrioventricular block;
* Killip >Ⅱ;
* Suspected acute myocardial infarction with heart rate<45 beats/min, P- R interval>0.24 sec or systolic blood pressure <100 mmHg;
* Existing contraindication for metoprolol or allergic to metoprolol or any excipients;
* Participation in another clinical study with an investigational product during the last 3 months;
* Previous enrolment in the present study;
* Subjects the investigator thinks not suitable for this study. E.g. cancer etc.;
* Inability to sign the informed consent form;
* Pregnancy or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
percentage of patients achieving target dose | 1 month
  The percentage of patients achieving target dose of 95mg/d at the time of discharge

SECONDARY OUTCOMES:
mean heart rate | 1 month
  The mean HR after achieving target dose
mean blood pressure | 1 month
  The mean BP after achieving target dose
percentage of patients who experienced bradycardia with symptoms | 1 month
  The percentage of patients who experienced bradycardia with symptoms during hospitalization and for 1 month after discharge, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, MD, Principal Investigator — The General Hospital of PLA
Locations (1):
- The General Hospital of PLA, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li D, Dong W, Liu Y, Wang J, Mu Y, Zhou H, Wang J, Zhou S, Chen Y. Impact of metoprolol standard dosing pathway in Chinese patients with acute coronary syndrome: protocol for a multicentre prospective study. BMJ Open. 2019 Dec 4;9(12):e031972. doi: 10.1136/bmjopen-2019-031972. PMID 31806613